CLINICAL TRIAL: NCT06548854
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Dose Exploration Clinical Trial Evaluating the Efficacy, Safety, and Pharmacokinetic Characteristics of STC314 Injection Administered Intravenously in Sepsis Patients
Acronym: Sepsis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grand Medical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPHIP-0203
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
Keywords: sepsis
MeSH Terms: conditions — Sepsis | interventions — STC3141

STUDY DESIGN:
Intervention Model Description: Three parallel groups were set up in this trial, including two different doses of STC314 injection treatment group (group 1 and group 2) and one placebo Dose control group (group 3).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study used 0.9% sodium chloride injection without any active drug as a placebo control, which was comparable to the characteristics and appearance of the experimental drug Imitation. The investigational drug and placebo are packaged and coded by a third party independent of the investigator and cannot be directly distinguished. by IWRS assigns study medication to subjects. Before database locking, subjects, researchers, in addition to DSMB and independent statistical teams and sponsors (including subjects and families, study physicians, study nurses, clinical coordinators, monitors, data managers, and statisticians) all were blind to the allocation of investigational drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose group (Experimental): The experimental drug was administered intravenously for 5 days
  Interventions: Drug: STC314 Injection/STC314 Injection Placebo
- low dose group (Experimental): The experimental drug was administered intravenously for 5 days
  Interventions: Drug: STC314 Injection/STC314 Injection Placebo
- Placebo (Placebo Comparator): Placebo infusion continued for 5 days
  Interventions: Drug: STC314 Injection/STC314 Injection Placebo

INTERVENTIONS:
Drug: STC314 Injection/STC314 Injection Placebo — All subjects who meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned to receive continuous intravenous infusion of STC314 injection (dose in salt form) or placebo with continuous intravenous infusion of the same volume load infusion for 5 days at an overall ratio of 1:1:1.
  Other Names: STC314 Injection Placebo

SUMMARY:
One study evaluated the efficacy and safety of intravenous STC314 injection in patients with sepsis Sex and pharmacokinetic profiles of a multicenter, randomized, double-blind, placebo-controlled II Phase I dose exploration clinical trial

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase II dose exploration study. The aim of this trial is to evaluate the efficacy, safety, and pharmacokinetic characteristics of STC314 injection in sepsis patients receiving loading dose and continuous intravenous infusion, determine the optimal therapeutic dose, and provide supporting evidence for phase III clinical trials. The overall design of the experiment is shown in Figure 1. This experiment consists of three parallel groups, including two treatment groups with different doses of STC314 injection and one placebo control group.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18≤ age ≤80 years old, gender is not limited; (2) The subjects or their guardians voluntarily participate in the study and sign the informed consent; (3) being treated in an intensive care unit; (4) Meet the diagnostic criteria for sepsis 3.0, namely:

  1. There is a confirmed or suspected infection;
  2. The presence of infection-induced organ dysfunction, i.e., the Sequential Organ failure score (SOFA) ≥2, as known in If there is organ function impairment before infection, that is, SOFA score is greater than 0, it is necessary to compare SOFA score after infection Previous rise ≥2 points. (5) SOFA score ≤ 13 points; (6) The time from meeting the sepsis 3.0 diagnostic criteria to randomization does not exceed 48 hours; (7) Male and female subjects of reproductive age agreed to use an effective contraceptive method from the start of the study until 1 month after the end of dosing.

Exclusion Criteria:

* (1) The pregnancy test of women of childbearing age before administration is positive, and pregnant or lactating women; (2) Chronic disease has caused serious organ function impairment, or has caused serious complications:

  1. Heart: New York Heart Association Heart Function Grade IV;
  2. Lung: chronic respiratory failure requires long-term oxygen therapy;
  3. Kidney: chronic kidney disease stage 4 or 5;
  4. Liver: previous liver failure, hepatic encephalopathy or hepatic coma, gastrointestinal bleeding caused by portal hypertension in the past six months; Or Child-Pugh score ≥ 10 points. (3) Cancer patients with cachexia, or due to obstruction, space occupation, extrusion and other reasons, resulting in serious damage to organ function or internal bleeding, Those who have difficulty or have not yet undergone surgical treatment, or who have received chemotherapy or immunotherapy within the last month; (4) The subjects had severe immune deficiency or were using strong immunosuppression: granulocytosis (N<0.5×10^9/L), activity Blood tumor or stage III HIV infection; Are being treated with immune-inducing drugs such as anti-thymocyte globulin (ATG), Antilymphocyte globulin (ALG), interleukin-2 receptor a chain antibody (IL-2RA), and interleukin-6 receptor αantibody (IL-6RA), etc. Continuous use of glucocorticoid therapy for nearly 2 weeks with a daily dose exceeding 200mg equivalent to hydrocortisone; (5) There is active bleeding that is difficult to control effectively; (6) Currently requiring systemic administration of therapeutic doses of anticoagulants (except prophylactic doses); (7) aPTT > 1.5 times the upper limit of normal value; (8) Platelet count < 50 ×10^9/L; (9) The patient needs or is receiving extracorporeal membrane oxygenation (ECMO) treatment; (10) endangered status, the expected survival time is not more than 24 hours; (11) Cardiac arrest, acute myocardial infarction, or massive cerebral infarction in the past 1 week; (12) are receiving or require dialysis or kidney replacement treatment within 6 hours; (13) Combined with severe or more severe burns: the total surface area of the burn exceeds 30% or the area of the third-degree burn exceeds 10%; Or surface Less than 30% of the volume, but the body condition is heavier or have shock, compound injury, respiratory tract burning; (14) Allergic to the active ingredient of the test drug (methylcellobiose sulfate) or excipients (disodium hydrogen phosphate and sodium dihydrogen phosphate); (15) Participants had participated in another clinical study (except those who did not receive intervention) or were participating in another trial within 1 month prior to screening Clinical treatment; (16) The subject's previous or ongoing disease, physical examination or laboratory test results are abnormal, as determined by the investigator to be probable Adversely affect the subject's safety in the study, or may affect the assessment of the subject's clinical or mental state By a wide margin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in sequential organ failure (SOFA) scores from baseline on day 7 value | 7 days after the first dose
  Changes in sequential organ failure (SOFA) scores from baseline on day 7 value

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wu, PM, Study Director — GrandPharma (China) Co., Ltd.
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China